CLINICAL TRIAL: NCT00453674
Title: Deutsches Nebennieren-Karzinom-Register - German Adrenocortical Carcinoma Registry
Brief Title: German Adrenocortical Carcinoma Registry
Status: Recruiting | Type: Observational
Sponsor: University of Wuerzburg (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Martin Fassnacht, Head of Endocrinology, University of Wuerzburg
Other Study IDs: Wue-ACC-R-86-03
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenal cancer; Treatment; Surgery; Mitotane
MeSH Terms: conditions — Adrenocortical Carcinoma; Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adrenocortical carcinoma: Adrenocortical carcinoma

SUMMARY:
Basic objective of the German Adrenocortical Carcinoma Registry is to improve the care of patients with adrenocortical cancer. The registration of as many patients as possible helps to collect data for the prognosis and prospects of success regarding different treatment plans. This data will be taken into consideration for planning prospective studies. With this registry, the recruitment of patients for prospective studies will be significantly facilitated. In this way - and in cooperation with networks in other countries (e.g. in Italy and France) - a structure allowing systematic improvement of therapy will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adrenocortical carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adrenocortical carcinoma patients in Germany (or treated in Germany)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2003-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fassnacht, MD, Principal Investigator — University of Wuerzburg
Locations (1):
- University of Wuerzburg, Würzburg, Germany

REFERENCES:
- [Result] Petersenn S, Richter PA, Broemel T, Ritter CO, Deutschbein T, Beil FU, Allolio B, Fassnacht M; German ACC Study Group. Computed tomography criteria for discrimination of adrenal adenomas and adrenocortical carcinomas: analysis of the German ACC registry. Eur J Endocrinol. 2015 Apr;172(4):415-22. doi: 10.1530/EJE-14-0916. Epub 2015 Jan 19. PMID 25599706
- [Result] Beuschlein F, Weigel J, Saeger W, Kroiss M, Wild V, Daffara F, Libe R, Ardito A, Al Ghuzlan A, Quinkler M, Osswald A, Ronchi CL, de Krijger R, Feelders RA, Waldmann J, Willenberg HS, Deutschbein T, Stell A, Reincke M, Papotti M, Baudin E, Tissier F, Haak HR, Loli P, Terzolo M, Allolio B, Muller HH, Fassnacht M. Major prognostic role of Ki67 in localized adrenocortical carcinoma after complete resection. J Clin Endocrinol Metab. 2015 Mar;100(3):841-9. doi: 10.1210/jc.2014-3182. Epub 2015 Jan 5. PMID 25559399
- [Result] Erdogan I, Deutschbein T, Jurowich C, Kroiss M, Ronchi C, Quinkler M, Waldmann J, Willenberg HS, Beuschlein F, Fottner C, Klose S, Heidemeier A, Brix D, Fenske W, Hahner S, Reibetanz J, Allolio B, Fassnacht M; German Adrenocortical Carcinoma Study Group. The role of surgery in the management of recurrent adrenocortical carcinoma. J Clin Endocrinol Metab. 2013 Jan;98(1):181-91. doi: 10.1210/jc.2012-2559. Epub 2012 Nov 12. PMID 23150691
- [Result] Hahner S, Kreissl MC, Fassnacht M, Haenscheid H, Knoedler P, Lang K, Buck AK, Reiners C, Allolio B, Schirbel A. [131I]iodometomidate for targeted radionuclide therapy of advanced adrenocortical carcinoma. J Clin Endocrinol Metab. 2012 Mar;97(3):914-22. doi: 10.1210/jc.2011-2765. Epub 2011 Dec 14. PMID 22170726
- [Result] Herrmann LJ, Heinze B, Fassnacht M, Willenberg HS, Quinkler M, Reisch N, Zink M, Allolio B, Hahner S. TP53 germline mutations in adult patients with adrenocortical carcinoma. J Clin Endocrinol Metab. 2012 Mar;97(3):E476-85. doi: 10.1210/jc.2011-1982. Epub 2011 Dec 14. PMID 22170717
- [Result] Reibetanz J, Jurowich C, Erdogan I, Nies C, Rayes N, Dralle H, Behrend M, Allolio B, Fassnacht M; German ACC study group. Impact of lymphadenectomy on the oncologic outcome of patients with adrenocortical carcinoma. Ann Surg. 2012 Feb;255(2):363-9. doi: 10.1097/SLA.0b013e3182367ac3. PMID 22143204
- [Result] Johanssen S, Hahner S, Saeger W, Quinkler M, Beuschlein F, Dralle H, Haaf M, Kroiss M, Jurowich C, Langer P, Oelkers W, Spahn M, Willenberg HS, Mader U, Allolio B, Fassnacht M. Deficits in the management of patients with adrenocortical carcinoma in Germany. Dtsch Arztebl Int. 2010 Dec;107(50):885-91. doi: 10.3238/arztebl.2010.0885. Epub 2010 Dec 17. PMID 21246024
- [Result] Fassnacht M, Johanssen S, Fenske W, Weismann D, Agha A, Beuschlein F, Fuhrer D, Jurowich C, Quinkler M, Petersenn S, Spahn M, Hahner S, Allolio B; German ACC Registry Group. Improved survival in patients with stage II adrenocortical carcinoma followed up prospectively by specialized centers. J Clin Endocrinol Metab. 2010 Nov;95(11):4925-32. doi: 10.1210/jc.2010-0803. Epub 2010 Jul 28. PMID 20668036
- [Result] Brix D, Allolio B, Fenske W, Agha A, Dralle H, Jurowich C, Langer P, Mussack T, Nies C, Riedmiller H, Spahn M, Weismann D, Hahner S, Fassnacht M; German Adrenocortical Carcinoma Registry Group. Laparoscopic versus open adrenalectomy for adrenocortical carcinoma: surgical and oncologic outcome in 152 patients. Eur Urol. 2010 Oct;58(4):609-15. doi: 10.1016/j.eururo.2010.06.024. Epub 2010 Jun 22. PMID 20580485
- [Result] Fassnacht M, Johanssen S, Quinkler M, Bucsky P, Willenberg HS, Beuschlein F, Terzolo M, Mueller HH, Hahner S, Allolio B; German Adrenocortical Carcinoma Registry Group; European Network for the Study of Adrenal Tumors. Limited prognostic value of the 2004 International Union Against Cancer staging classification for adrenocortical carcinoma: proposal for a Revised TNM Classification. Cancer. 2009 Jan 15;115(2):243-50. doi: 10.1002/cncr.24030. PMID 19025987
- [Result] Quinkler M, Hahner S, Wortmann S, Johanssen S, Adam P, Ritter C, Strasburger C, Allolio B, Fassnacht M. Treatment of advanced adrenocortical carcinoma with erlotinib plus gemcitabine. J Clin Endocrinol Metab. 2008 Jun;93(6):2057-62. doi: 10.1210/jc.2007-2564. Epub 2008 Mar 11. PMID 18334586
- [Result] Terzolo M, Angeli A, Fassnacht M, Daffara F, Tauchmanova L, Conton PA, Rossetto R, Buci L, Sperone P, Grossrubatscher E, Reimondo G, Bollito E, Papotti M, Saeger W, Hahner S, Koschker AC, Arvat E, Ambrosi B, Loli P, Lombardi G, Mannelli M, Bruzzi P, Mantero F, Allolio B, Dogliotti L, Berruti A. Adjuvant mitotane treatment for adrenocortical carcinoma. N Engl J Med. 2007 Jun 7;356(23):2372-80. doi: 10.1056/NEJMoa063360. PMID 17554118
- [Result] Fassnacht M, Hahner S, Polat B, Koschker AC, Kenn W, Flentje M, Allolio B. Efficacy of adjuvant radiotherapy of the tumor bed on local recurrence of adrenocortical carcinoma. J Clin Endocrinol Metab. 2006 Nov;91(11):4501-4. doi: 10.1210/jc.2006-1007. Epub 2006 Aug 8. PMID 16895957
- [Result] Kimpel O, Bedrose S, Megerle F, Berruti A, Terzolo M, Kroiss M, Mai K, Dekkers OM, Habra MA, Fassnacht M. Adjuvant platinum-based chemotherapy in radically resected adrenocortical carcinoma: a cohort study. Br J Cancer. 2021 Oct;125(9):1233-1238. doi: 10.1038/s41416-021-01513-8. Epub 2021 Aug 16. PMID 34400803
- [Result] Kimpel O, Schindler P, Schmidt-Pennington L, Altieri B, Megerle F, Haak H, Pittaway J, Dischinger U, Quinkler M, Mai K, Kroiss M, Polat B, Fassnacht M. Efficacy and safety of radiation therapy in advanced adrenocortical carcinoma. Br J Cancer. 2023 Feb;128(4):586-593. doi: 10.1038/s41416-022-02082-0. Epub 2022 Dec 8. PMID 36482186
- [Result] Kroiss M, Megerle F, Kurlbaum M, Zimmermann S, Wendler J, Jimenez C, Lapa C, Quinkler M, Scherf-Clavel O, Habra MA, Fassnacht M. Objective Response and Prolonged Disease Control of Advanced Adrenocortical Carcinoma with Cabozantinib. J Clin Endocrinol Metab. 2020 May 1;105(5):1461-8. doi: 10.1210/clinem/dgz318. PMID 31900481
- [Result] Reibetanz J, Rinn B, Kunz AS, Flemming S, Ronchi CL, Kroiss M, Deutschbein T, Pulzer A, Hahner S, Kocot A, Germer CT, Fassnacht M, Jurowich C. Patterns of Lymph Node Recurrence in Adrenocortical Carcinoma: Possible Implications for Primary Surgical Treatment. Ann Surg Oncol. 2019 Feb;26(2):531-538. doi: 10.1245/s10434-018-6999-z. Epub 2018 Nov 15. PMID 30443830
- [Result] Megerle F, Herrmann W, Schloetelburg W, Ronchi CL, Pulzer A, Quinkler M, Beuschlein F, Hahner S, Kroiss M, Fassnacht M; German ACC Study Group. Mitotane Monotherapy in Patients With Advanced Adrenocortical Carcinoma. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1686-1695. doi: 10.1210/jc.2017-02591. PMID 29452402
- [Result] Henning JEK, Deutschbein T, Altieri B, Steinhauer S, Kircher S, Sbiera S, Wild V, Schlotelburg W, Kroiss M, Perotti P, Rosenwald A, Berruti A, Fassnacht M, Ronchi CL. Gemcitabine-Based Chemotherapy in Adrenocortical Carcinoma: A Multicenter Study of Efficacy and Predictive Factors. J Clin Endocrinol Metab. 2017 Nov 1;102(11):4323-4332. doi: 10.1210/jc.2017-01624. PMID 29092062
- See also: Official website of the German Adrenocortical Carcinoma Study Group — https://www.nebennierenkarzinom.de/
- See also: Homepage of the Dept. of Endocrinology Wuerzburg — https://www.ukw.de/medizinische-klinik-i/endokrinologie/startseite/